CLINICAL TRIAL: NCT04009291
Title: PaTH Forward: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Trial With an Open-Label Extension, Investigating the Safety, Tolerability and Efficacy of TransCon PTH Administered Subcutaneously Daily in Adults With Hypoparathyroidism
Brief Title: A Trial Investigating the Safety, Tolerability and Efficacy of TransCon PTH in Adults With Hypoparathyroidism
Acronym: PaTH Forward
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TransCon PTH TCP-201
Expanded Access: NCT05654701 (Approved for marketing)
Record Dates: First submitted 2019-06-20; First posted 2019-07-05 (Actual); Results first posted 2023-09-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Hypoparathyroidism; Endocrine System Diseases; Parathyroid Diseases
Keywords: Hypoparathyroidism; Parathyroid Hormone; PTH(1-34); Prodrug; Sustained Release; TransCon PTH; Parathyroid Hormone Replacement Therapy
MeSH Terms: conditions — Hypoparathyroidism; Endocrine System Diseases; Parathyroid Diseases

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled, parallel group with subjects randomized into 4 treatment groups (1:1:1:1): Transcon PTH 15 mcg/day, TransCon PTH 18 mcg/day, TransCon PTH 21 mcg/day, placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TransCon PTH 15 mcg (Experimental): TransCon PTH 15 mcg delivered once daily by subcutaneous injection
  Interventions: Combination Product: TransCon PTH
- TransCon PTH 18 mcg (Experimental): TransCon PTH 18 mcg delivered once daily by subcutaneous injection
  Interventions: Combination Product: TransCon PTH
- TransCon PTH 21 mcg (Experimental): TransCon PTH 21 mcg delivered once daily by subcutaneous injection
  Interventions: Combination Product: TransCon PTH
- Placebo (Placebo Comparator): Placebo mimicking 15, 18, or 21 mcg of TransCon PTH delivered once daily by subcutaneous injection
  Interventions: Combination Product: Placebo for TransCon PTH
- Open-Label Extension Period (Experimental): Subjects who complete the four-week blinded period are assigned to open-label treatment with TransCon PTH for up to 262 weeks, with up to an initial 14 weeks of TransCon PTH titration and standard of care optimization, followed by approximately 248 weeks of individualized dosing.
  Interventions: Combination Product: TransCon PTH

INTERVENTIONS:
Combination Product: TransCon PTH — TransCon PTH drug product is supplied as a clear solution containing TransCon PTH with a nominal PTH(1-34) content of 0.3 mg/mL in a pre-filled pen intended for subcutaneous injection.
  Arms: Open-Label Extension Period; TransCon PTH 15 mcg; TransCon PTH 18 mcg; TransCon PTH 21 mcg
Combination Product: Placebo for TransCon PTH — Placebo is supplied as a clear solution containing the formulation buffer for TransCon PTH in a pre-filled pen intended for subcutaneous injection.
  Arms: Placebo

SUMMARY:
During the first four weeks of the trial, participants will be randomly assigned to one of four groups: three groups will receive fixed doses of TransCon PTH and one group will receive placebo. TransCon PTH or placebo will be administered as a subcutaneous injection using a pre-filled injection pen. Neither trial participants nor their doctors will know who has been assigned to each group. After the four weeks, participants will continue in the trial as part of a long-term extension study. During the extension, all participants will receive TransCon PTH, with the dose adjusted to their individual needs. This is a global trial that will be conducted in, but not limited to, the United States, Canada, Germany, Denmark, and Norway.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥18 years.
2. Subjects with postsurgical chronic HP or auto-immune, genetic, or idiopathic HP for at least 26 weeks.
3. On a stable dose for at least 12 weeks (or 4 weeks if on Natpara as of September 2019) prior to Screening of:

   * ≥0.25 μg BID of calcitriol (active vitamin D) or ≥0.5 μg BID or ≥1.0 μg daily of alfacalcidol (active vitamin D), and
   * ≥400 mg BID calcium citrate or carbonate.
4. Optimization of supplements prior to randomization to achieve the target levels of:

   * 25(OH) vitamin D levels of 30-70 ng/mL (75-175 pmol/mL) and
   * Magnesium level within the normal range and
   * Albumin-adjusted or ionized serum calcium (sCa) level in the lower half of the normal range.
5. BMI 17-40 kg/m2 at Visit 1.
6. If ≤25 years of age, radiological evidence of epiphyseal closure based on x-ray of non-dominant wrist and hand.
7. eGFR >30 mL/min/1.73m2 during Screening.
8. Thyroid-stimulating hormone (TSH) within normal laboratory limits within the 12 weeks prior to Visit 1; if on suppressive therapy for thyroid cancer, TSH level must be ≥0.2 μIU/mL.
9. If treated with thyroid hormone replacement therapy, the dose must be stable for at least 12 weeks prior to Visit 1.
10. Able to perform daily subcutaneous self-injections of study drug (or have a designee perform injection) via a pre-filled injection pen.
11. Written, signed, informed consent of the subject.

Exclusion Criteria:

1. Known activating mutation in the calcium-sensing receptor (CaSR) gene.
2. Impaired responsiveness to PTH (pseudohypoparathyroidism) which is characterized as PTH-resistance, with elevated PTH Levels in the setting of hypocalcemia.
3. Any disease that might affect calcium metabolism or calcium-phosphate homeostasis or PTH levels other than HP, such as active hyperthyroidism; Paget's disease; hypomagnesemia; type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus; severe and chronic cardiac, liver, or renal disease; Cushing syndrome; rheumatoid arthritis; multiple myeloma; active pancreatitis; malnutrition; rickets; recent prolonged immobility; active malignancy (other than low-risk well differentiated thyroid cancer or basal cell skin cancer); parathyroid carcinoma within 5 years prior to Screening; acromegaly; multiple endocrine neoplasia types 1 and 2.
4. Use of loop diuretics, phosphate binders (other than calcium carbonate/calcium citrate), digoxin, lithium, methotrexate, or systemic corticosteroids (other than replacement therapy).
5. Use of thiazide diuretic within 4 weeks prior to the Screening 24-hour urine collection or the first dose adjustment of SOC during Screening.
6. Use of PTH-like drugs (whether commercially available or through participation in an investigational trial) including PTH(1-84), PTH(1-34), or other N-terminal fragments or analogs of PTH or PTH-related protein within 5 weeks prior to Visit 1.
7. Use of other drugs known to influence calcium and bone metabolism, such as calcitonin, fluoride tablets (> 0.5 mg/day), strontium, or cinacalcet hydrochloride within 12 weeks prior to Visit 1.
8. Use of bisphosphonates (oral or IV) or denosumab within 2 years prior to Visit 1.
9. Non-hypocalcemic seizure disorder with a history of a seizure within 26 weeks prior to Visit 1.
10. Increased risk for osteosarcoma, such as those with Paget's disease of bone or unexplained elevations of alkaline phosphatase, open epiphyses, hereditary disorders predisposing to osteosarcoma, or with a prior history of substantial external beam or implant radiation therapy involving the skeleton.
11. Pregnant or lactating women. Note: Highly effective contraception (see Appendix 7) is required for sexually active women of childbearing potential during the trial and for 2 weeks after the last dose of study drug, and pregnancy testing will be performed throughout the trial. Sexually active women of childbearing potential who are unwilling to use highly effective contraception are excluded from the trial.
12. Diagnosis of drug or alcohol dependence within 3 years prior to Visit 1.
13. Disease processes that may adversely affect gastrointestinal absorption including but not limited to short bowel syndrome, bowel resection, gastric bypass, tropical sprue, active celiac disease, active ulcerative colitis, gastroparesis, AIRE gene mutations with malabsorption, and active Crohn's disease.
14. Chronic or severe cardiac disease within 26 weeks prior to Visit 1 including but not limited to congestive heart failure, myocardial infarction, QTcF >430 msec (males) or >450 msec (females), severe or uncontrolled arrhythmias, bradycardia (resting heart rate <50 beats/minute), symptomatic hypotension, systolic BP <80 mm Hg or diastolic <40 mm Hg, or poorly controlled hypertension (systolic BP >150 mm Hg or diastolic >95 mm Hg).
15. Cerebrovascular accident within 5 years prior to Visit 1.
16. History of renal colic or acute gout within 52 weeks prior to Visit 1.
17. Any disease or condition that, in the opinion of the investigator, may make the subject unlikely to fully complete the trial, or any condition that presents undue risk from the investigational product or procedures, including treated malignancies that are likely to recur within the approximate 1-year duration of the trial.
18. Known allergy or sensitivity to PTH or any of the excipients.
19. Participation in another clinical trial in which receipt of investigational drug or device occurred within 8 weeks (or at least 5.5 times the half-life of the investigational drug) prior to Visit 1.
20. Likely to be non-compliant with respect to trial conduct.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2025-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Shu, MD, Study Director — Ascendis Pharma A/S Medical Monitor/Medical Expert
Locations (15):
- United States (5):
  - Ascendis Pharma Investigational Site, Chicago, Illinois
  - Ascendis Pharma Investigational Site, Rochester, Minnesota
  - Ascendis Pharma Investigational Site, Great Neck, New York
  - Ascendis Pharma Investigational Site, New York, New York
  - Ascendis Pharma Investigational Site, Philadelphia, Pennsylvania
- Ascendis Pharma Investigational Site, Oakville, Ontario, Canada
- Denmark (3):
  - Ascendis Pharma Investigational Site, Aalborg
  - Ascendis Pharma Investigational Site, Aarhus
  - Ascendis Pharma Investigational Site, Copenhagen
- Ascendis Pharma Investigational Site, Dresden, Germany
- Italy (4):
  - Ascendis Pharma Investigational Site, Bologna
  - Ascendis Pharma Investigational Site, Milan
  - Ascendis Pharma Investigational Site, Pisa
  - Ascendis Pharma Investigational Site, Rome
- Ascendis Pharma Investigational Site, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khan AA, Rejnmark L, Rubin M, Schwarz P, Vokes T, Clarke B, Ahmed I, Hofbauer L, Marcocci C, Pagotto U, Palermo A, Eriksen E, Brod M, Markova D, Smith A, Pihl S, Mourya S, Karpf DB, Shu AD. PaTH Forward: A Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial of TransCon PTH in Adult Hypoparathyroidism. J Clin Endocrinol Metab. 2022 Jan 1;107(1):e372-e385. doi: 10.1210/clinem/dgab577. PMID 34347093
- [Derived] Khan AA, Rubin MR, Schwarz P, Vokes T, Shoback DM, Gagnon C, Palermo A, Marcocci C, Clarke BL, Abbott LG, Hofbauer LC, Kohlmeier L, Pihl S, An X, Eng WF, Smith AR, Ukena J, Sibley CT, Shu AD, Rejnmark L. Efficacy and Safety of Parathyroid Hormone Replacement With TransCon PTH in Hypoparathyroidism: 26-Week Results From the Phase 3 PaTHway Trial. J Bone Miner Res. 2023 Jan;38(1):14-25. doi: 10.1002/jbmr.4726. Epub 2022 Nov 12. PMID 36271471

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 104 subjects were screened and 59 of these met eligibility criteria and were enrolled into the study. The four-week blinded period is completed and the study is ongoing with all participants receiving TransCon PTH in the open-label period.
Groups:
- Open-Label TransCon PTH: Subjects who completed the four-week blinded period were assigned to open-label treatment with TransCon PTH for up to 262 weeks, with up to an initial 14 weeks of TransCon PTH titration and standard of care optimization, followed by approximately 248 weeks of individualized dosing.
Period: Blinded Period (Weeks 0 to 4)
Arm/Group | TransCon PTH 15 mcg | TransCon PTH 18 mcg | TransCon PTH 21 mcg | Placebo | Open-Label TransCon PTH
Started | 14 | 15 | 15 | 15 | 0
Completed | 14 | 15 | 15 | 15 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Open-Label Period (Weeks 4 to 266)
Arm/Group | TransCon PTH 15 mcg | TransCon PTH 18 mcg | TransCon PTH 21 mcg | Placebo | Open-Label TransCon PTH
Started | 0 | 0 | 0 | 0 | 59
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 59
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Study Ongoing | 0 | 0 | 0 | 0 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TransCon PTH 15 mcg | TransCon PTH 18 mcg | TransCon PTH 21 mcg | Placebo | Total
Number analyzed (Participants) | 14 | 15 | 15 | 15 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.03 (13.230) | 46.58 (11.157) | 53.67 (11.287) | 51.80 (12.345) | 49.82 (12.094)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 12 | 12 | 48
  Male | 2 | 3 | 3 | 3 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 15 | 14 | 15 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 2 | 0 | 2
  White | 14 | 12 | 13 | 15 | 54
  Other | 0 | 3 | 0 | 0 | 3
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] | 166.92 (8.806) | 166.71 (8.385) | 165.37 (10.961) | 164.07 (10.368) | 165.75 (9.520)
Weight [Mean (Standard Deviation); unit: kg] | 76.58 (22.479) | 80.04 (11.279) | 72.26 (18.621) | 76.43 (14.256) | 76.32 (16.869)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.08 (5.723) | 28.76 (3.148) | 26.12 (4.647) | 28.30 (3.775) | 27.57 (4.415)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - Primary Endpoint During the Blinded Period
Description: The percentage of subjects with albumin-adjusted serum calcium within the normal range, and spot morning fractional excretion of calcium (spot AM FECa) within normal range (≤2%) or a reduction by at least 50% from baseline, and not taking active vitamin D supplements, and taking ≤1000 mg/day of calcium supplements
Time Frame: Week 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TransCon PTH 15 mcg | TransCon PTH 18 mcg | TransCon PTH 21 mcg | Placebo
Number analyzed (Participants) | 14 | 15 | 15 | 15
Percentage of participants | 50.0 [23.0 to 77.0] | 40.0 [16.3 to 67.7] | 60.0 [32.3 to 83.7] | 26.7 [7.8 to 55.1]
Statistical Analysis 1: Comparison: TransCon PTH 15 mcg vs Placebo; Fisher's exact test is used to compare differences in the proportion of subjects meeting the composite primary endpoint in the TransCon PTH versus pooled placebo group; Test type: Superiority; p = 0.2635, t-test, 2 sided
Statistical Analysis 2: Comparison: TransCon PTH 18 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6999, t-test, 2 sided
Statistical Analysis 3: Comparison: TransCon PTH 21 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1394, t-test, 2 sided

2. Secondary Outcome: Efficacy - Key Secondary Endpoint During the Blinded Period
Description: The percentage of subjects with albumin-adjusted serum calcium within the normal range, and spot AM FECa within the normal range (≤2%) or a reduction by at least 50% from baseline, and not taking active vitamin D supplements, and taking ≤ 500 mg/day of calcium supplements
Time Frame: Week 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TransCon PTH 15 mcg | TransCon PTH 18 mcg | TransCon PTH 21 mcg | Placebo
Number analyzed (Participants) | 14 | 15 | 15 | 15
Percentage of participants | 50.0 [23.0 to 77.0] | 26.7 [7.8 to 55.1] | 60.0 [32.3 to 83.7] | 20.0 [4.3 to 48.1]
Statistical Analysis 1: Comparison: TransCon PTH 15 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1281, t-test, 2 sided
Statistical Analysis 2: Comparison: TransCon PTH 18 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p > 0.9999, t-test, 2 sided
Statistical Analysis 3: Comparison: TransCon PTH 21 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0604, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 Week Blinded Period and Open-Label Period starting at Week 4 up to Week 84
Groups:
- TransCon PTH Period: The total period of exposure to TransCon PTH. For subjects randomized to TransCon PTH at enrollment, this was the time from the first dose of blinded TransCon PTH until data cutoff in the open-label extension (OLE) period. The TransCon PTH Period for subjects randomized to placebo at enrollment was the time from first exposure to TransCon PTH at the time of cross-over from placebo, until data cutoff in the OLE.
Arm/Group | TransCon PTH 15 mcg | TransCon PTH 18 mcg | TransCon PTH 21 mcg | Placebo | TransCon PTH Period
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/15 | 0/15 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/15 | 0/15 | 5/59
Other Adverse Events (participants affected / at risk) | 6/14 | 5/15 | 7/15 | 6/15 | 51/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TransCon PTH 15 mcg (N=14) | TransCon PTH 18 mcg (N=15) | TransCon PTH 21 mcg (N=15) | Placebo (N=15) | TransCon PTH Period (N=59)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papillary tumour of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3.4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TransCon PTH 15 mcg (N=14) | TransCon PTH 18 mcg (N=15) | TransCon PTH 21 mcg (N=15) | Placebo (N=15) | TransCon PTH Period (N=59)
Headache (Nervous system disorders) | 3 | 1 | 1 | 1 | 13
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 4
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 6
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 4
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 7
Injection site pain (General disorders) | 1 | 0 | 1 | 0 | 2
Thirst (General disorders) | 0 | 1 | 1 | 0 | 2
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 6
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 7
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 5
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 4
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 2
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Keratitis (Eye disorders) | 0 | 0 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 2
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 2
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT04009291/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT04009291/SAP_002.pdf